CLINICAL TRIAL: NCT04310306
Title: First-pass Recanalization With EmboTrap II in Acute Ischemic Stroke (FREE-AIS)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2019-1057
Record Dates: First submitted 2020-03-13; First posted 2020-03-17 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Acute Ischemic Stroke Due to Intracranial Large Artery Occlusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Rescue stenting group
  Interventions: Device: Thrombectomy using EmboTrap II

INTERVENTIONS:
Device: Thrombectomy using EmboTrap II — The subjects will receive endovascular treatment for acute stroke according to standard clinical practice. Specifically, using a stent retriever, contact aspiration EmboTrap II. The number of thrombectomy attempts is at the operator's discretion. Combination of balloon guide catheter or intermediate catheter is recommended.

SUMMARY:
This study is a prospective, open-label, multi-center, registry study, designed to to documents that EmboTrap II usage as a thrombectomy device for emergency large vessel occlusion (ELVO) in terms of the rate of First Pass Recanalization (FPR). Patients with ELVO will initially underwent mechanical thrombectomy usig EmboTrap II. FPR is defined as modified Tissue Thrombolysis In Cerebral Ischemia (mTICI) 2b or 3

ELIGIBILITY:
Inclusion Criteria:

1. Subjects experiencing acute ischemic stroke due to large vessel occlusion (intracranial internal carotid artery and middle cerebral artery M1 or proximal M2 segment, intracranial vertebral artery and basilar artery
2. Age 19 or greater
3. mRS before qualifying stroke, 0 to 2
4. Baseline NIHSS score 4 or more
5. CT ASPECTS > 5 or MR ASPECTS > 4
6. Good collateral statues on CT angiogram (collateral grade by Calgary group, 4 or 5) or corresponding to DEFUSE 3 or DAWN trial on perfusion imaging.
7. Onset (last-seen-well) time to femoral puncture time < 24 hours
8. Anticipated life expectancy of at least 12 months
9. Patients who undergo endovascular thrombectomy with EmboTrap II as the first-line device
10. Signed informed consent for study enrollment

Exclusion Criteria:

1. Multiple simultaneous large vessel occlusions
2. Pregnancy
3. Severe contrast allergy or absolute contraindication to iodinated contrast agent
4. Patient has a severe or fatal combined illness that will prevent improvement of follow-up or will render the procedure unlikely to benefit the patient.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute stroke due to ELVO within 24 hours after last seen well
Sampling Method: Non-Probability Sample
Enrollment: 310 (Estimated)
Dates: Start 2020-02-10 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
First Pass Recanalization (FPR) rate | Within 1 day after the completion of endovascular thrombectomyh
  The rate of FPR defined by modified TICI 2b or 3

SECONDARY OUTCOMES:
The rate of modified Rankin scale 0-2 at 3 months after treatment | 90 days ± 14 days
  The rate of modified Rankin Scale score (mRS), 0-2 at 90 days ± 14 days

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital Stroke Center, Yonsei University College of Medicine, Seongdu, South Korea

IPD SHARING:
Plan to Share IPD: Undecided